CLINICAL TRIAL: NCT00032435
Title: CSP #453 - Homocysteinemia in Kidney and Endstage Renal Disease Study (HOST)
Brief Title: Homocysteine Study (HOST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Pan American Laboratories (Industry); Abbott Diagnostics Division (Industry)
Responsible Party: Jamison, Rex - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Masking: Double
Other Study IDs: 453
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: End Stage Renal Disease; Renal Failure
Keywords: folate; pyridoxine; vitamin B6; cyanocobalamin; homoc
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PAL-40 Active
  Interventions: Drug: PAL-40 Active
- 2 (Placebo Comparator): PAL-40 Placebo
  Interventions: Drug: PAL-40 Placebo

INTERVENTIONS:
Drug: PAL-40 Active
  Arms: 1
Drug: PAL-40 Placebo
  Arms: 2

SUMMARY:
The primary objective of this study is to test the hypothesis that administration of folate, pyridoxine (vitamin B6) and cyanocobalamin (vitamin B12) in high doses to patients with advanced chronic renal failure or end stage renal disease and abnormally high plasma homocysteine levels will lower the homocysteine levels and the death rate compared to patients who receive placebo. The secondary objective is to test the hypothesis that intake of the vitamins compared to placebo decreases the incidence of myocardial infarction, disabling stroke, and amputation of a lower extremity and, in hemodialysis patients, thrombosis of the vascular access.

DETAILED DESCRIPTION:
Primary Hypothesis:

The primary objective of this proposal is to test the hypothesis that administration of folate, pyridoxine (vitamin B6) and cyanocobalamin (vitamin B12) in high doses to patients with advanced chronic renal failure or end-stage renal disease and abnormally high plasma homocysteine levels will lower the homocysteine levels and increase survival.

Secondary Hypotheses:

The secondary objectives are to test the hypotheses that intake of the vitamins decreases: 1) MI, 2) stroke, 3) amputation of lower extremity, 4) combination death, MI, stroke and amputation of lower extremity, 5) thrombosis of the vascular access in hemodialysis patients.

Primary Outcome: Death

Interventions: A treated group that receives a daily tablet containing 40mg of folic acid, 100mg of pyridoxine and 2mg of B12 versus a control group that receives a placebo.

Study Abstract:

The experimental design is a prospective, two-arm, randomized, double blind study, stratified for medical center and whether the patient has chronic renal failure or end-stage renal disease. In each arm 1003 patients will ingest daily a capsule containing either 40mg of folic acid, 100mg of pyridoxine and 2mg of vitamin B12, or placebo. We will use stratified randomization to ensure that the treatment is balanced within the end-stage renal disease patients and chronic renal failure patients.

This 6 year study will require an accrual phase of 2 years and a treatment phase lasting a minimum of 4 years. Patients will be screened by their plasma homocysteine concentration. They must have a level of at least 15 uM/L to be enrolled in the study. The study nurse will evaluate each patient at 3 months. Thereafter, patients will be contacted by phone, or mail if they prefer, at 3-month intervals by coordinators at a central location. Secondary endpoint events, hospitalization, onset of dialysis, and death or other reason for exit from the study will be recorded on standard forms. Plasma homocysteine levels will be obtained at 3 months in all patients.

Patients will be excluded if: age less than 21 years, expected life span less than 6 months, pregnancy, metastatic cancer, AIDS-related infection, end-stage liver disease, vitamin B12 deficiency, treatment with methotrexate, or anticonvulsants, unreliable or likely non-compliant, participation in other long-term trial, or unwilling or unable to give informed consent.

For a relative treatment effect of 17% (that is reducing the 3-year death rate from 28% to 23.2%) and 80% power, 2006 patients and 36 VA medical centers are required.

An abundance of published reports has shown a strong correlation between homocysteinemia and the incidence of cardiovascular death. Authors of these papers have unanimously recommended a study be undertaken to determine if folate, pyridoxine, and vitamin B12 can lower the incidence.

The study is to be conducted in patients with chronic renal failure and end-stage renal disease whose plasma homocysteine levels and incidence of cardiovascular death and disease are among the highest of all patient populations. By screening for patients with high plasma homocysteine concentrations and measuring the levels after 3 months, we will be able to determine if the hypothetical reduction in death and cardiovascular event rate is associated with a decrease in plasma homocysteine concentration.

ELIGIBILITY:
Inclusion Criteria:

Patients will be screened by their plasma homocysteine concentration. They must have a level of at least 15 mM/L to be enrolled in the study.

Patients will be excluded by any of the following criteria: age less than 21 years, expected life span less than 6 months, pregnancy, metastatic cancer, end-stage liver disease, treatment with methotrexate, other anti-folate medication or anticonvulsants, unreliable or likely noncompliant, participation in another long-term trial, or unwilling or unable to give informed consent.

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2003 (Estimated)
Dates: Start 2001-05; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rex L. Jamison, Study Chair — VA Palo Alto Health Care System
Locations (37):
- United States (36):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Health Economics Resource Center (HERC), Menlo Park, Menlo Park, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Medical Center, Miami, Miami, Florida
  - West Palm Beach VA Medical Center, West Palm Beach, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - Southeast Veterans Healthcare System, New Orleans, New Orleans, Louisiana
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, Jackson, Mississippi
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Northport, Northport, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - VA Medical Center, Bronx, The Bronx, New York
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Dayton, Dayton, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Derived] Brady CB, Gaziano JM, Cxypoliski RA, Guarino PD, Kaufman JS, Warren SR, Hartigan P, Goldfarb DS, Jamison RL. Homocysteine lowering and cognition in CKD: the Veterans Affairs homocysteine study. Am J Kidney Dis. 2009 Sep;54(3):440-9. doi: 10.1053/j.ajkd.2009.05.013. Epub 2009 Jul 23. PMID 19628319
- [Derived] Jamison RL, Shih MC, Humphries DE, Guarino PD, Kaufman JS, Goldfarb DS, Warren SR, Gaziano JM, Lavori P; Veterans Affairs Site Investigators. Effect of the MTHFR C677T and A1298C polymorphisms on survival in patients with advanced CKD and ESRD: a prospective study. Am J Kidney Dis. 2009 May;53(5):779-89. doi: 10.1053/j.ajkd.2008.12.023. Epub 2009 Mar 9. PMID 19272686
- [Derived] Jamison RL, Hartigan P, Kaufman JS, Goldfarb DS, Warren SR, Guarino PD, Gaziano JM; Veterans Affairs Site Investigators. Effect of homocysteine lowering on mortality and vascular disease in advanced chronic kidney disease and end-stage renal disease: a randomized controlled trial. JAMA. 2007 Sep 12;298(10):1163-70. doi: 10.1001/jama.298.10.1163. PMID 17848650